CLINICAL TRIAL: NCT05019079
Title: Protective Effect of Electroacupuncture on Lung in Patients Undergoing General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lingling Ding (Other)
Responsible Party: Sponsor-Investigator, Lingling Ding, Professor, Beijing Hospital of Traditional Chinese Medicine
Organization: Beijing Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LDing
Record Dates: First submitted 2021-07-25; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Electroacupuncture; Lung Injury, Ventilator Induced
Keywords: Electroacupuncture; Lung protection; ventilator induced lung injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture group (Experimental): In the electroacupuncture group, acupoints of Lieque (+), Chize (-), Sanyinjiao (-), Zusanli (+), Tanzhong (+) and Yutang (-) will be selected for electrical stimulation. Density wave will be selected, and the current intensity should be tolerated by the patients. Conventional anesthesia operation could be started after the connection of electroacupuncture, and acupuncture point stimulation was stopped 30min later.
  Interventions: Other: electroacupuncture
- control group (No Intervention): The patient underwent routine anesthesia without acupuncture treatment

INTERVENTIONS:
Other: electroacupuncture — In the electroacupuncture group, acupoints of Lieque (+), Chize (-), Sanyinjiao (-), Zusanli (+), Tanzhong (+) and Yutang (-) will be selected for electrical stimulation. Density wave will be selected, and the current intensity should be tolerated by the patients. Conventional anesthesia operation could be started after the connection of electroacupuncture, and acupuncture point stimulation will be stopped 30min later.
  Arms: electroacupuncture group

SUMMARY:
Objective to investigate the protective effect of preoperative electroacupuncture on lung function in patients with mechanical ventilation for more than 2 hours under general anesthesia

DETAILED DESCRIPTION:
Randomized parallel control study. From September 1, 2021 to December 31, 2022, patients with mechanical ventilation time more than 2 hours will be randomly divided into electroacupuncture pretreatment group and blank control group. The blood gas index, ventilator parameters and serum inflammatory factor concentration of patients will be evaluated to evaluate whether electroacupuncture has protective effect on lung function of patients with mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia in our hospital;
* Ages 18-60;
* American Society of Anesthesiologists (ASA) grade ⅱ ~ III , no severe respiratory, circulation, liver, kidney, coagulation function abnormalities;
* Expected duration of operation >2h;
* Surgical grade 2-4;
* No serious lung infection and lung disease;
* Body mass index (BMI) 18~30 kg/m2; There are no contraindications for electroacupuncture stimulation.

Exclusion Criteria:

* Patients with severe circulatory or other system dysfunction;
* Patients with pulmonary and one-lung ventilation;
* Unwilling to cooperate with the patient;
* Patients with low compliance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
oxygenation index | Before anesthesia
  record oxygenation index
oxygenation index | 2 hours after tracheal intubation
  record oxygenation index
oxygenation index | 5 minutes after tracheal intubation removal
  record oxygenation index

SECONDARY OUTCOMES:
Postoperative comfort score | during anesthesia recovery period
  Assess the quality of recovery during recovery
sedation score (Ramsay) | during anesthesia recovery period
  Assess the quality of recovery during recovery
restfulness score (DRS) | during anesthesia recovery period
  Assess the quality of recovery during recovery
visual analogue scale (VAS) | during anesthesia recovery period
  Assess the quality of recovery during recovery
Length of stay | 1 week after discharge, the patient's length of stay will be recorded through medical record system
  Assess the quality of postoperative recovery
postoperative time in hospital | 1 week after discharge, the patient's postoperative time in hospital will be recorded through medical record system
  Assess the quality of postoperative recovery
postoperative complications of major organs | Major organ complications during hospitalization，assessed up to 30 days after surgery
  Assess the quality of postoperative recovery
mortality within 30 days | mortality within 30 days will be recorded
  Assess the quality of postoperative recovery
Expression of IL-18 in serum | Before anesthetic induction the radial artery blood samples will be collected, and the expressions of IL-18 in serum will be detected by flow cytometry
  The perioperative inflammation level will be assessed
Expression of IL-18 in serum | 5minutes after tracheal intubation removal the radial artery blood samples will be collected, and the expressions of IL-18 in serum will be detected by flow cytometry
  The perioperative inflammation level will be assessed
Expression of IL-1β in serum | Before anesthetic induction the radial artery blood samples will be collected, and the expressions of IL-1β in serum will be detected by flow cytometry
  The perioperative inflammation level will be assessed
Expression of IL-1β in serum | 5minutes after tracheal intubation removal the radial artery blood samples will be collected, and the expressions of IL-1β in serum will be detected by flow cytometry
  The perioperative inflammation level will be assessed
Expression of IL-10 in serum | Before anesthetic induction the radial artery blood samples will be collected, and the expressions of IL-10 in serum will be detected by flow cytometry
  The perioperative inflammation level will be assessed
Expression of IL-10 in serum | 5minutes after tracheal intubation removal the radial artery blood samples will be collected, and the expressions of IL-10 in serum will be detected by flow cytometry
  The perioperative inflammation level will be assessed
Mean arterial pressure | Before anesthesia ,2 hours after tracheal intubation , and 5minutes after tracheal intubation removal
  Intraoperative vital signs will be recorded
heart rate | Before anesthesia , 2 hours after tracheal intubation , and 5minutes after tracheal intubation removal
  Intraoperative vital signs will be recorded
BIS | Before anesthesia , 2 hours after tracheal intubation , and 5minutes after tracheal intubation removal
  Intraoperative vital signs will be recorded
extubation time | Before anesthesia , 2 hours after tracheal intubation , and 5minutes after tracheal intubation removal
  Intraoperative vital signs will be recorded
anesthesia dosage | Before anesthesia , 2 hours after tracheal intubation , and 5minutes after tracheal intubation removal
  Intraoperative vital signs will be recorded